CLINICAL TRIAL: NCT02748577
Title: Pain Processing in Adults With Migraines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00027845
Record Dates: First submitted 2016-04-11; First posted 2016-04-22 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2019-08

CONDITIONS: Migraines
Keywords: Migraines; Pain responses
MeSH Terms: conditions — Migraine Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Migraine (Experimental): Participants with migraines will complete one study visit where they will complete several questionnaires and will also complete Quantitative Sensory Testing (QST) Pain Measurements. They must be migraine-free during the visit and no migraine within 48 hrs of study visit
  Interventions: Other: Questionnaires; Other: Quantitative Sensory Testing (QST) Pain Measurements
- Healthy Controls (Active Comparator): Healthy Controls will complete one study visit where they will complete several questionnaires and will complete Quantitative Sensory Testing (QST) Pain Measurements.
  Interventions: Other: Questionnaires; Other: Quantitative Sensory Testing (QST) Pain Measurements

INTERVENTIONS:
Other: Questionnaires — Before the experimental session, participants will use REDCap to complete several questionnaires used to assess outcomes.
Other: Quantitative Sensory Testing (QST) Pain Measurements — Investigators will administer noxious thermal stimulation to assess pain threshold temperatures and assess responses to pain on measures of pain intensity and pain unpleasantness

SUMMARY:
Primary Objective of this study: To assess experimental heat pain responses (pain intensity, pain unpleasantness, pain catastrophizing, emotional reactivity) in migraineurs vs. healthy controls.

The current tools of migraine pain measurement are inadequate to distinguish the overall burden of suffering, as there is an over reliance on a single numerical pain score to represent the entire pain experience. Measuring and targeting the affective component, in addition to the sensory component of pain, may capture this discrepancy in disease burden. The affective component of migraine pain may be just as important as the sensory component to target and measure since it significantly impacts outcomes, disability, and has therapeutic treatment implications.

Quantitative sensory testing (QST) is a robust lab paradigm (not a clinical experience) that delivers one painful noxious thermal stimuli and asks for simultaneous pain intensity and pain unpleasantness scores. By using this in the research, investigators will be able to differentiate the sensory (pain quality-what the pain feels like) from the affective (how awful/unpleasant the pain feels) components of experimental pain in normal controls vs. migrainuers.

No previous studies have evaluated differences in experimental pain intensity vs. pain unpleasantness in migraineurs vs. controls. As migraine pain uniquely involves many altered sensory phenomenon (e.g., photophobia, phonophobia), it cannot be assumed that responses to experimental pain in migraine will be the same as other clinical pain syndromes. Further, different clinical pain syndromes have distinct responses to pain intensity vs. pain unpleasantness.

DETAILED DESCRIPTION:
Investigators will conduct a cross-sectional study in migraineurs (interictally, i.e., between migraine attacks) and healthy controls to compare responses to experimental heat pain intensity and unpleasantness and correlate these results to differences in emotional reactivity and pain catastrophizing.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for Healthy Controls:

   * ≥18yo;
2. Inclusion Criteria for Migraineurs:

   * ≥18yo with >1 yr of migraines and currently 4-20 days/month with migraines, although no migraine within 48 hrs of study visit.

Exclusion Criteria:

1. Any major unstable medical/psychiatric illness (e.g., hospitalization within 90 days, suicide risk, etc.)
2. Severe clinical depression/anxiety
3. Chronic pain condition (e.g., fibromyalgia, migraines for healthy controls, etc.) or sensory abnormalities (e.g., neuropathy, Raynaud's, etc.)
4. Diagnosis of medication overuse headache or chronic migraine.
5. Migraineurs will be studied after being headache-free for at least 48 hours (interictally).
6. Participants may be currently taking migraine medications, as long as they do not have a diagnosis of medication overuse headache.
7. Pregnant subjects will be excluded from all portions of the study due to possible unknown risks of frankly noxious stimuli.
8. Due to unknown risks and potential harm to the unborn fetus, sexually active women of childbearing potential must use a reliable method of birth control while participating in this study
9. Volunteers with no pain ratings to frankly noxious stimuli (temperatures > 49°C) or excessive responses to threshold temperatures (~43°C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Heat Pain Intensity coefficient and intercept from stimulus response curve | One visit
  Using the logarithmic equation: log (VAS pain ratings)=log (t - 35) * coefficient + intercept where t represents stimulus temperature, we will generate stimulus-response curves for each subject
Heat Pain Unpleasantness coefficient and intercept from stimulus response curve | One visit
  Using the logarithmic equation: log (VAS pain ratings)=log (t - 35) * coefficient + intercept where t represents stimulus temperature, we will generate stimulus-response curves for each subject
Pain Catastophizing score | One Visit
  Score on the Pain Catastrophizing instrument
Difficulty in Emotions Regulation score | One Visit
  Score on the Difficulty in Emotions Regulation score

SECONDARY OUTCOMES:
Heat Pain Threshold Temperature | One Visit
  Temperature of heat pain threshold
Anxiety | One Visit
  Score on the Generalized Anxiety Disorder (GAD-7) instrument
Depression | One Visit
  Score on the Patient Health related questionnaire-depression module (PHQ-9) instrument
Mindfulness | One Visit
  Score on the Five Factor Mindfulness (FFM) instrument
Stress | One Visit
  Score on the Perceived Stress Scale (PSS) instrument
Hope | One Visit
  Score on the Herth Hope Index instrument
Optimism | One Visit
  Score on the Life Orientation Test instrument
Social Connectedness | One Visit
  Score on the Social Connectedness Scale instrument
Flourishing | One Visit
  Score on the Flourishing scale instrument
Resilience | One Visit
  Score on the Brief Resilience scale instrument
Sleep | One Visit
  Score on the NIH Promis Measure of sleep disturbance instrument
Global Health | One Visit
  Score on the 1st question of the NIH Promis Global Health measure

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Wells, MD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Access Criteria: Please contact the study principal investigator, Dr. Rebecca Wells rewells@wakehealth.edu, for the study protocol and other information

DOCUMENTS (1):
  • Informed Consent Form (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT02748577/ICF_000.pdf